CLINICAL TRIAL: NCT04675008
Title: A Phase II Study of Dacomitinib in Advanced Epidermal Growth Factor Receptor (EGFR)-Mutant Non-small Cell Lung Cancer (NSCLC) Patients Who Have Non-irradiated Brain Metastasis
Brief Title: Central Nervous System(CNS) Efficacy of Dacomitinib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong-Mu Sun, Associated Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2020-09-117
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Non Small Cell Lung Cancer; Brain Metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Dacomitinib
  Interventions: Drug: Dacomitinib

INTERVENTIONS:
Drug: Dacomitinib — Secondary generation EGFR-tyrosine kinase inhibitor (TKI) (Dacomitinib) for EGFR mutant NSCLC patients with non irradiated brain metastasis
  Other Names: Vizimpro

SUMMARY:
This is a single-arm, phase II study of dacomitinib in advanced EGFR-mutant NSCLC patients who have non-irradiated brain metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven recurrent or metastatic NSCLC (adenocarcinoma) with major EGFR mutation (exon 19 deletion or Leu858Arg mutation without the Thr790Met)
* No prior systemic treatment of advanced NSCLC (Neoadjuvant or adjuvant chemotherapy are allowed, without limitation on its treatment timing)
* Age ≥20 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Had at least one measurable intracranial lesion as ≥ 5mm in the longest diameter by magnetic resonance imaging (MRI) (≥ 5mm by thin section (1.2mm) of brain MRI image, ≥ 10mm by less thin section(2.5mm) brain MRI ), which checked within 4 weeks before enrollment. If MRI slice thickness is not appropriate, we need to recheck Brain MRI
* Number of brain metastasis =>5
* Adequate organ function
* Female subjects must either be of non-reproductive potential
* Subject is willing and able to comply with the protocol
* Signed written informed consent

Exclusion Criteria:

* Severe symptomatic brain metastasis, needing urgent control with radiotherapy or high dose steroid: the definition of high dose steroid is the equivalent dose of dexamethasone 10 mg or higher per day (mild symptoms controlled with low dose of steroid can be enrolled)
* With leptomeningeal seeding
* Exposure to EGFR-TKIs or other EGFR targeting agents at any time in either neoadjuvant or adjuvant setting
* Local treatment (stereotatic radiosurgery or whole brain radiotherapy) for brain metastases
* Uncontrolled systemic illness including uncontrolled hypertension, active bleeding, or active infection.
* Past medical history of interstitial lung disease, drug induced interstitial lung disease, radiation pneumonitis which required steroid treatment
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-07 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
CNS objective response rate (Complete response or Partial response) | 1 year
  The rate of CR or PR of CNS disease

SECONDARY OUTCOMES:
CNS progression-free survival | 1 year
  Time from enrollment to CNS progression or death
Cumulative incidence of CNS failure by competing risk analysis | 1 year
  To evaluate the CNS efficacy of dacomitinib
Extracranial objective response rate | 1 year
  The rate of CR or PR
Progression-free survival | 1 year
  Time from enrollment to progression or death
Overall survival | 1 year
  Time from enrollment to death of any cause
Safety by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 1 year
  The % of side effect

CONTACTS AND LOCATIONS:
Locations (1):
- Jong-Mu Sun, Seoul, South Korea